CLINICAL TRIAL: NCT00844974
Title: Cognitive Deficits in Major Depressive Disorder and Bipolar Disorder Depressed Type: Prevalence and Symptoms With Treating of Depressive Symptoms
Brief Title: Cognitive Deficits in Major Depressive Disorder and Bipolar Disorder, Depressed Type: Prevalence and Improvement With Treatment of Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John D. Matthews, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2007-p-001665
Record Dates: First submitted 2008-05-08; First posted 2009-02-16 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Major Depression; Bipolar Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Prevalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Other: Prevalence

INTERVENTIONS:
Other: Prevalence — Mood and cognitive assessments

SUMMARY:
The purpose of this research study is to learn more about cognitive deficits in people with certain mood disorders. The mood disorders are Major Depressive Disorder (MDD) and Bipolar disorder, depressed type.

Cognitive deficits are problems with things like thinking and memory. People with cognitive deficits may have problems concentrating and paying attention. When talking, they may have trouble recalling a word they want to say. They may think slowly and have problems remembering things. These deficits can affect an individual's ability to work and function socially. Cognitive deficits that occur with depression may increase the risk of a relapse of major depressive disorder.

We want to study the course of cognitive impairment in subjects as they are receiving treatment for their depression. We want to find out if their cognitive deficits get better, worse, or stay the same.

We also want to learn more about a stress hormone called cortisol that is produced in the body. We want to study the relationship between cortisol and cognitive impairment. Recent research has shown that cognitive impairment may be more severe in people who have high levels of cortisol in their blood.

We will also measure the levels of a protein in your blood called brain-derived neurotrophic factor (BDNF). BDNF helps the growth of new brain cells. It appears that the growth of new brain cells lessens when people are depressed. Treatment with antidepressant medications may cause BDNF levels to increase and return to normal. We are interested in studying the relationship between BDNF levels and cognitive impairment throughout treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible subjects will be inpatients admitted to the Massachusetts General Psychiatric inpatient service, Blake 11 with diagnoses of MDD with and without psychotic features and BPDD with and without psychotic features.
2. Subjects will include men and women aged 18-85.
3. Competent to give informed consent.

Exclusion Criteria:

1. Patients with illnesses that impair cognitive functioning including: vascular dementia, and neurological illnesses including Parkinson's Disease, Huntington's Disease, multiple sclerosis, and Alzheimer's Disease.
2. The following DSM-IV diagnoses: schizophrenia, schizoaffective disorder, delusional disorder, organic mental disorder, substance use disorders including alcohol, active within the past 6 months, acute bereavement, and psychotic disorder not elsewhere classified.
3. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To examine the relationship between severity and type of depression with cognitive deficits | study duration

CONTACTS AND LOCATIONS:
Overall Officials: John D Matthews, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States